CLINICAL TRIAL: NCT04585373
Title: Time Course Effects of Kinesio-taping in Knee Osteoarthritis Patients.
Brief Title: Effects of Kinesio-taping in Knee Osteoarthritis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00679 Anila kausar
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis
Keywords: kinseotaping; Osteoarthritis; Degenerative joint; Numeric pain rating scale; Time up and go test; Functional reach test; Western Ontario osteoarthritis index
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (24 hours) (Experimental): kinesio-tapping along with conventional therapy
  Interventions: Other: kinesio-taping with conventional therapy 24 hours
- (48hours) (Experimental): kinesio-tapping along with conventional therapy
  Interventions: Other: kinesio-taping with conventional therapy 48 hours
- (72 hours) (Experimental): kinesio-tapping along with conventional therapy
  Interventions: Other: kinesio-taping with conventional therapy 72 hours

INTERVENTIONS:
Other: kinesio-taping with conventional therapy 24 hours — standardized therapeutic KT application along with conventional therapy (hot pack ,strengthening and stretching exercises) quadriceps tapping: In the supine position, the Y shape tape will be applied from the middle of the thigh to the upper edge of the patella, Then, the tape will anchored to the inner and outer aspect of the patella with 25% muscle tension and the distal end of the strips are positioned on the tibial tubercle without any tension.
  McConnell Patellar tapping technique:
  The patient will be positioned in long sitting position; affected knee joint exposed. As per McConnell patellar taping technique, tape will applied from superior and lateral patellar borders, maximally pulling it medially. A second strip can be used for reinforcement, but it should not cover the popliteal fossa.
  Arms: (24 hours)
Other: kinesio-taping with conventional therapy 48 hours — standardized therapeutic KT application along with conventional therapy (hot pack ,strengthening and stretching exercises) quadriceps tapping: In the supine position, the Y shape tape will be applied from the middle of the thigh to the upper edge of the patella, Then, the tape will anchored to the inner and outer aspect of the patella with 25% muscle tension and the distal end of the strips are positioned on the tibial tubercle without any tension.
  McConnell Patellar tapping technique:
  The patient will be positioned in long sitting position; position; affected knee joint exposed. As per McConnell patellar taping technique, tape will applied from superior and lateral patellar borders, maximally pulling it medially. A second strip can be used for reinforcement, but it should not cover the popliteal fossa.
  Arms: (48hours)
Other: kinesio-taping with conventional therapy 72 hours — standardized therapeutic KT application along with conventional therapy (hot pack ,strengthening and stretching exercises) quadriceps tapping: In the supine position, the Y shape tape will be applied from the middle of the thigh to the upper edge of the patella, Then, the tape will anchored to the inner and outer aspect of the patella with 25% muscle tension and the distal end of the strips are positioned on the tibial tubercle without any tension.
  McConnell Patellar tapping technique:
  The patient will be positioned in long sitting position; affected knee joint exposed. As per McConnell patellar taping technique, tape will applied from superior and lateral patellar borders, maximally pulling it medially. A second strip can be used for reinforcement, but it should not cover the popliteal fossa.
  Arms: (72 hours)

SUMMARY:
The main reason to conduct this research is to find the comparison of kinseotaping according to time duration that is 24 hours, 48 hours and 72 hours in knee osteoarthritis patients. We can find the impact of kinseo-taping on pain, balance and functional status of patients.

DETAILED DESCRIPTION:
Osteoarthritis is a common, slowly developing disease which is enhance with age, it is also called as metabolic disease, which includes destruction and repair mechanisms that begin by bio chemical and mechanical injury. Knee osteoarthritis is a chronic degenerative disease. Because of aging and due to obesity and sedentary lifestyle risk factor in prevalence of knee osteoarthritis is increased. Cartilage is the main tissue affected by osteoarthritis and causes following symptoms including pain, stiffness, joint swelling and also decrease the range of motion. It is the one of main cause of deformity which results in poor quality of life. Knee osteoarthritis is most occurring from all types of joint disease. The WHO estimated that Osteoarthritis will become the fourth main cause of disability the year 2020. Knee pain may affect knee flexibility and cause functional disability. Quadriceps muscle weakness is one of the most marked disability impairment that is seen in knee osteoarthritis patients. This linked to functional limitations which increase fall risk and slower walking speed.

Muscle strength test showed that knee osteoarthritis patient have 25% to 45% loss of knee extension strength and 19% to 25% loss of knee flexion strength. The prevalence and incidence of knee osteoarthritis is greater in patient with age 30-65 years then adults population. Approximately 80% patients of knee osteoarthritis experience from movement restriction and 20% are not able to perform daily living activates and 11% experience from personal care. In developed countries knee osteoarthritis affects 17% to 30% of elderly population over age of 65 years and more prevalence in women than men. It is evaluate that by 2020 the approximately number of people diagnosed with osteoarthritis will be 57% and those individuals whose is affected by movement limitation will be approximately 66% Osteoarthritis is most prevalent form of joint arthritis. Knee osteoarthritis accounts for pain and functional disability in 19.2-27.8% of people age >45, approximately 37%of individual age >60 had knee osteoarthritis in plain radiography. Knee osteoarthritis is 4.9%over age 26 years, 16.7% among individual over 45 years and 12.1% over age 60 years. Osteoarthritis is rheumatologic disease which affects 80% of individual above 55 years. The current world wide prevalence of knee osteoarthritis is 3.8% and women are affected more often 4.8% then men. In united state knee osteoarthritis prevalence's increases by 66-100% by 2020. The main goal of knee osteoarthritis treatment is to decrease pain and maintain loss of physical function.

Among other conservative techniques use in knee osteoarthritis patients, the use of different kind of taping approaches for treatment of knee osteoarthritis patients. Kinseotaping was described use in clinics for pain management and motor function enhancement in patients of musculoskeletal injuries. Kinseotaping improve muscle flexibility and muscle strength it also improve proprioception in patients of musculoskeletal symptoms. It has been shown that elastic tape could increase local circulation, decrease edema, and maintain joint stability. Kinseotaping method is an alternative elastic taping techniques which is specially designed waterproof, hypo allergic elastic tape. This tape should apply directly on skin and left for several days. This tape would provide therapeutic effects.Kinseo-taping has high elastic adhesive material and also high stretching capacity to give free mobility at applied area. This kinseotaping improve knee pain by improving patellofemoral alignment and decrease mechanical stress on soft tissue. The kinseotaping is elastic woven cotton strip with heat sensitive acrylic adhesive and can stretch 120%-140% of its original length. It has been suggested that kinseotaping provide cutaneous stimulation which reduce pain by activating mechanoreceptors and improve muscle excitability Kinseotaping reverse the pain signals through stimulating sensory nerve endings of skin. It has been evaluated that taping on patella can improve patellar proprioception and sense of mechanical stability.

In 2019 study compares the effect of quadriceps taping with patellar taping to check balance and functional performance in patients of knee osteoarthritis. The result showed that both quadriceps and patellar taping equally improve balance and functional level of knee osteoarthritis patients. Another research was conducted in 2019in which they describe the immediate effects of kinseotaping on gait function and pain in older patients of knee osteoarthritis. Result showed that kinseotaping significantly improved gait and balance and it also decreased the pain during ambulation. In 2018 study evaluate the gait speed after applying kinseotaping on quadriceps femoris muscle in knee osteoarthritis patients. Their result suggest that time needed to perform 10 meter walk test would decreased after 3 days of application of kinseo-taping.In 2017study conducted research on effects of kinseotaping on pain and functional outcome in knee osteoarthritis patients ,their result revealed that therapeutic kinseotaping is effective in short term management of pain and disability in knee osteoarthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral and bilateral knee OA
* O.A with grade 2-3(Kellgren and Lawrence system for classification of osteoarthritis of knee)
* Experiencing Pain for more than 1 month

Exclusion Criteria:

* Rheumatic diseases, inflammatory arthritis, septic arthritis
* Intra-articular corticosteroid injection during the past month
* Patients with fracture
* Patients with any carcinoma
* if patient having any other systemic illness.
* Allergic reaction to KT

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 72 hour
  numeric pain rating scale is used to assess the intensity of pain before and after intervention. Its value ranges from 0-10. O indicates no pain and 10 indicate maximum pain. Reliability of this tool is r=0.957. It will be measured at 24 hour,48 hour,72 hour
Western Ontario and McMaster Universities Osteoarthritis index | 72 hour
  Western Ontario and McMaster Universities Osteoarthritis index is used to measure the primary outcomes of pain and physical function. This questionnaire includes 24 questions divided into 3 subscales pain, stiffness and physical function. f=0.39 . It will be measured at 24 hour,48 hour,72 hour
Time Up and Go | 72 hour
  time up and go test is used to assess the dynamic balance ability, in this subject took to rise from 46cm height arm chair, walk 3 meter, turn back at affected side and walk back to chair and sit. Reliability of this tool is r = 0.98 to 0.99. It will be measured at 24 hour,48 hour,72 hour
function reach test | 72 hour
  function reach test is used to measure the balance in this ask the patient to stand close to wall, position the arm at 90 degree of shoulder flexion. The therapist record location of 3 Metacarpal head. Ask the patient to reach as far as possible without taking a step. The location of 3rd MC Head recorded again. The difference between start and end position was Reach distance. Reliability is r=0.151. It will be measured at 24 hour,48 hour,72 hour

CONTACTS AND LOCATIONS:
Overall Officials: Shafaq Shahid, MSPT(OMPT), Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tani K, Kola I, Shpata V, Dhamaj F. Evaluation of Gait Speed after Applying Kinesio Tape on Quadriceps Femoris Muscle in Patients with Knee Osteoarthritis. Open Access Maced J Med Sci. 2018 Aug 15;6(8):1394-1398. doi: 10.3889/oamjms.2018.273. eCollection 2018 Aug 20. PMID 30159063
- [Background] Taheri P, Vahdatpour B, Asl MM, Ramezanian H. Effects of Taping on Pain and Functional Outcome of Patients with Knee Osteoarthritis: A Pilot Randomized Single-blind Clinical Trial. Adv Biomed Res. 2017 Nov 10;6:139. doi: 10.4103/2277-9175.218031. eCollection 2017. PMID 29279837
- [Background] Lu Z, Li X, Chen R, Guo C. Kinesio taping improves pain and function in patients with knee osteoarthritis: A meta-analysis of randomized controlled trials. Int J Surg. 2018 Nov;59:27-35. doi: 10.1016/j.ijsu.2018.09.015. Epub 2018 Sep 28. PMID 30273684
- [Background] Li X, Zhou X, Liu H, Chen N, Liang J, Yang X, Zhao G, Song Y, Du Q. Effects of Elastic Therapeutic Taping on Knee Osteoarthritis: A Systematic Review and Meta-analysis. Aging Dis. 2018 Apr 1;9(2):296-308. doi: 10.14336/AD.2017.0309. eCollection 2018 Apr. PMID 29896418
- [Background] Abolhasani M, Halabchi F, Afsharnia E, Moradi V, Ingle L, Shariat A, Hakakzadeh A. Effects of kinesiotaping on knee osteoarthritis: a literature review. J Exerc Rehabil. 2019 Aug 28;15(4):498-503. doi: 10.12965/jer.1938364.182. eCollection 2019 Aug. PMID 31523668
- [Background] Cho HY, Kim EH, Kim J, Yoon YW. Kinesio taping improves pain, range of motion, and proprioception in older patients with knee osteoarthritis: a randomized controlled trial. Am J Phys Med Rehabil. 2015 Mar;94(3):192-200. doi: 10.1097/PHM.0000000000000148. PMID 25706053
- [Background] Aydogdu O, Sari Z, Yurdalan SU, Polat MG. Clinical outcomes of kinesio taping applied in patients with knee osteoarthritis: A randomized controlled trial. J Back Musculoskelet Rehabil. 2017 Sep 22;30(5):1045-1051. doi: 10.3233/BMR-169622. PMID 28655128
- [Background] Park JS, Yoon T, Lee SH, Hwang NK, Lee JH, Jung YJ, Lee G. Immediate effects of kinesiology tape on the pain and gait function in older adults with knee osteoarthritis. Medicine (Baltimore). 2019 Nov;98(45):e17880. doi: 10.1097/MD.0000000000017880. PMID 31702659
- [Background] Donec V, Kubilius R. The effectiveness of Kinesio Taping(R) for pain management in knee osteoarthritis: a randomized, double-blind, controlled clinical trial. Ther Adv Musculoskelet Dis. 2019 Aug 29;11:1759720X19869135. doi: 10.1177/1759720X19869135. eCollection 2019. PMID 31497072
- [Background] Ouyang JH, Chang KH, Hsu WY, Cho YT, Liou TH, Lin YN. Non-elastic taping, but not elastic taping, provides benefits for patients with knee osteoarthritis: systemic review and meta-analysis. Clin Rehabil. 2018 Jan;32(1):3-17. doi: 10.1177/0269215517717307. Epub 2017 Jun 29. PMID 28660785
- [Background] Tani K, Kola I, Dhamaj F, Shpata V, Zallari K. Physiotherapy Effects in Gait Speed in Patients with Knee Osteoarthritis. Open Access Maced J Med Sci. 2018 Mar 10;6(3):493-497. doi: 10.3889/oamjms.2018.126. eCollection 2018 Mar 15. PMID 29610607
- [Background] Lee K, Yi CW, Lee S. The effects of kinesiology taping therapy on degenerative knee arthritis patients' pain, function, and joint range of motion. J Phys Ther Sci. 2016 Jan;28(1):63-6. doi: 10.1589/jpts.28.63. Epub 2016 Jan 30. PMID 26957729
- [Background] Rahlf AL, Braumann KM, Zech A. Kinesio Taping Improves Perceptions of Pain and Function of Patients With Knee Osteoarthritis: A Randomized, Controlled Trial. J Sport Rehabil. 2019 Jul 1;28(5):481-487. doi: 10.1123/jsr.2017-0306. Epub 2018 Dec 12. PMID 29466081
- [Background] Gomes CAFP, Dibai-Filho AV, Biasotto-Gonzalez DA, Politti F, Camillo de Carvalho PT. Association of Pain Catastrophizing With Static Balance, Mobility, or Functional Capacity in Patients With Knee Osteoarthritis: A Blind Cross-sectional Study. J Manipulative Physiol Ther. 2018 Jan;41(1):42-46. doi: 10.1016/j.jmpt.2017.08.002. Epub 2017 Dec 15. PMID 29249415